CLINICAL TRIAL: NCT06607328
Title: Comparison of Activity Restriction, Activity Performance Level, Kinesiophobia, Quality of Life, and Self-efficacy Levels of Prehypertensive and Hypertensive Individuals
Brief Title: Comparison of Prehypertensive and Hypertensive Individuals
Status: Completed | Type: Observational
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Betül Taşpınar, Study Director, Izmir Democracy University
Other Study IDs: HYPERTENSION-35
Record Dates: First submitted 2024-09-17; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Hypertension; Prehypertension
Keywords: Prehypertension; Hypertension; Limitation of activity; Occupational performance; Kinesiophobia; Quality of life; Self-efficacy
MeSH Terms: conditions — Hypertension; Prehypertension; Kinesiophobia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prehypertensive Group (PHTG): The prehypertensive group (PHTG) was formed from the prehypertensive individuals with similar characteristics.
  Interventions: Other: Assessment of participants in terms of different aspects.
- Hypertensive Group (HTG): In line with the Holter results hypertensive group (HTG) was formed from the individuals who were followed up with the diagnosis of hypertension.
  Interventions: Other: Assessment of participants in terms of different aspects.

INTERVENTIONS:
Other: Assessment of participants in terms of different aspects. — This group was composed of individuals who have the prehypertensive stage.

SUMMARY:
Blood pressure is a physiological indicator that occurs due to the change in the pressure exerted by the blood in the vessel during the systole and diastole of the heart, which has similar results among people. Multiple pathophysiological mechanisms can be responsible for elevated blood pressure. In this change, hypertension is defined as conditions in which blood pressure rises above normal values and the pressure generated in the vessel wall can be measured as a numerical (quantitative) value. Many factors can affect arterial blood pressure, morbidity, and mortality rates such as activity limitation, activity performance level, kinesiophobia, quality of life, self-efficacy levels, physical activity, and comorbidity levels. According to our knowledge, there are almost no studies comparing prehypertensive and hypertensive individuals in the literature, so it is important to create appropriate treatment programs by taking precautions in the early period. Therefore, this study aimed to compare activity limitation, activity performance level, kinesiophobia, quality of life, self-efficacy levels, physical activity, and comorbidity levels of prehypertensive and hypertensive individuals.

DETAILED DESCRIPTION:
Blood pressure (BP) is a physiological indicator that occurs due to the change in the pressure exerted by the blood in the vessel during the systole and diastole of the heart, which has similar results among people. The pressure exerted by the blood on the artery wall due to cardiac output and total peripheral resistance is called "arterial blood pressure". Multiple pathophysiological mechanisms can be responsible for elevated blood pressure. In this change, hypertension is defined as conditions in which blood pressure rises above normal values and the pressure generated in the vessel wall can be measured as a numerical (quantitative) value. Many factors can affect arterial blood pressure. Due to these factors, deviations in normal values of blood pressure may occur. While expressing the relationship between high blood pressure and physical activity, the Turkish Society of Cardiology states that individuals with sedentary life habits are more likely to have hypertension by 20-50% compared to those who regularly engage in physical activity. The guideline of the American Joint Committee for the National Assembly emphasizes that keeping blood pressure below 140/90 mmHg values during the HT process will reduce morbidity and mortality rates. The high Charlson comorbidity index results of individuals show that it is associated with high morbidity and mortality rates. Studies have shown that kinesiophobia, which is seen among the causes of high blood pressure in individuals, is associated with musculoskeletal pain, low back pain, fibromyalgia, and coronary artery diseases. Since the decrease in the level of activity is related to the fear of moving, it may be thought that blood pressure may increase in individuals if fear and anxiety are repeated. There is a relationship between activity limitation and age, and individuals over the age of 75 experience limitations in activities, there are studies that show a significant difference between hypertension and activity limitation between individuals who use anti-hypertensive drugs and individuals who do not, as well as studies in which contrary results are reported. Increasing the awareness of individuals about healthy living behaviors greatly impacts the control and follow-up of diseases in the disease process, as well as improving their self-efficacy while undertaking their health responsibilities, thus protecting their health. To make healthy living behaviors a habit, raising awareness of individuals about behavior change processes and what kind of result they can achieve when they do what action they do helps them to increase their self-effectiveness, and it is important to maintain and include them in daily life habits as well as increasing self-effectiveness. Quality of life is a concept determined by individuals' subjective perception and the interaction of physical, psychological, social, and environmental factors. Beyond the health status of the individual, this concept also encompasses his experiences in a wide range of life, functional capacity, mental health, social relations, and environmental interactions. In the literature, it is stated that individuals' physical habits, levels, limitations, personal beliefs, fear of moving, activity performance, and satisfaction are related to their quality of life. There is no study in the literature on the activity performance of hypertensive individuals, so it is thought that our study will make important contributions at the national and international levels. As a result, there are almost no studies comparing prehypertensive and hypertensive individuals in the literature, so it is important to create appropriate treatment programs by taking precautions in the early period. Therefore, this study aimed to compare activity limitation, activity performance level, kinesiophobia, quality of life, self-efficacy levels, physical activity, and comorbidity levels of prehypertensive and hypertensive individuals.

ELIGIBILITY:
Inclusion Criteria:

Criteria for inclusion for HTG;

* Age range is between 18 and 65 years
* According to blood pressure holter records, 24-hour average blood pressure values are SBP ≥139 mmHg and DBB ≥89 mmHg and hypertension diagnosis record
* Not having an orthopedic problem that prevents walking
* Volunteering to participate in research

Criteria for inclusion for PHTG;

* Age range is between 18 and 65 years
* According to blood pressure holter records, 24-hour average blood pressure values should be in the range of 120-139 mmHg for SBP and 80-89 mmHg for DBB
* Not having an orthopedic problem that prevents walking
* Volunteering to participate in research

Exclusion Criteria:

The exclusion criteria for HTG;

* To be diagnosed with a cerebral tumor, degenerative neurological diseases, epilepsy, or mental retardation that cause communication problems
* Loss of consciousness due to head trauma
* Having a history of pathology or fracture involving the lower extremity in the last six months

Exclusion criteria for PHTG;

* To be diagnosed with a cerebral tumor, degenerative neurological diseases, epilepsy, or mental retardation that cause communication problems
* Loss of consciousness due to head trauma
* Having a history of pathology or fracture involving the lower extremity in the last six months

Ages: 22 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study was conducted with individuals with prehypertension and hypertension who were followed up with Holter at M. Akif Ersoy Cardiovascular Surgery Hospital. An informed consent form was obtained from the participants who met the inclusion criteria and volunteered to participate in the study after being informed about the scope of the research. In line with the Holter results, the hypertensive group (HTG) was formed from the individuals who were followed up with the diagnosis of hypertension, and the prehypertensive group (PHTG) was formed from the prehypertensive individuals with similar characteristics.
Sampling Method: Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Assessment of Activity Limitation | 12 month
  Activity limitation was evaluated with Groningen Activity Restriction Scale. It consists of 18 items that score the degree of ability to perform daily routine life habits from 1 to 5 points. A minimum of 18x1:18 points and 18x5:90 points can be obtained from this measurement tool. A score of 18 indicates that there is no disability and a score of 90 indicates an advanced disability.
Assessment of Kinesiophobia | 12 month
  To measure kinesiophobia, Tampa Kinesiophobia Rating for Heart (CTKD) measurement tool was used in the study. The scale consists of a total of 17 items, including fear of injury, avoidance of exercise, perceived danger for heart problems, and dysfunction sub-dimensions. The level of kinesiophobia increases as the total score obtained from the measurement tool, which can be obtained with a minimum of 17 points and a maximum of 68 points, increases.
Assessment of Quality of Life | 12 month
  The MacNew Health-Related Quality of Life Questionnaire, which is applied in heart disease, was used to measure quality of life (QOL) in prehypertensive and hypertensive individuals. The measurement tool was created with 27 items in a seven-point Likert type. To measure the level of QOL in individuals with heart disease, each item can be scored from one to seven. This scale is divided into three sub-dimensions: physical, emotional, and social, and a total score can be obtained between 27 and 189. It was stated that the higher the total scores, the higher the QOL, while it was stated that the QOL level decreased as the score level decreased
Assessment of Self-efficacy | 12 month
  The self-efficacy assessment of prehypertensive and hypertensive individuals was evaluated with the Hypertension Self-Efficacy Scale. This scale consists of 20 items. Each item of the measurement tool is given a score between one and four for the options not suitable at all, not suitable, suitable, and very suitable. A total of a minimum of 20 to a maximum of 80 points can be obtained from the scale. It is stated that as the total score increases in individuals with high blood pressure, the level of self-efficacy also increases, that is, the degree of compliance with the treatment protocol increases
Assessment of Physical Activity | 12 month
  Physical activity levels of hypertensive and prehypertensive individuals, the International Physical Activity Questionnaire Short Form was used. Questions are used to determine the amount of time spent walking, sitting, and moderate and vigorous activities. As a result of calculations, the total physical activity score is found by adding the scores expressed in the three categories to each other. Physical activity levels are evaluated by determining these inactive, moderately active, and very active.
Assessment of Comorbidity Level | 12 month
  The Charlson Comorbidity Index is a scoring system that includes 19 comorbidity diagnoses. The measurement tool evaluates the mortality risk of comorbidities between one and six points. In the comorbidity index, which is scored according to the morbidity and mortality of the diseases, dementia, myocardial infarction, congestive heart failure, ulcer disease, cerebrovascular, peripheral vascular diseases, chronic pulmonary disease, connective tissue disease, diabetes mellitus, mild liver diseases are scored as "1 point". In the presence of leukemia, hemiplegia, moderate or severe renal diseases, malignant lymphoma, diabetes mellitus with end-organ damage, malignancy, "2 points" are scored. The sum of all measurement tool scores constitutes the CKI index's total score. I
Assessment of Activity Performance | 12 month
  The Canadian Activity Performance Scale was used. In the measurement tool, individuals are asked about their productivity, leisure activities and the degree to which they can and cannot care for themselves, that is, performance measurements. Individuals determine the five activities themselves in order of importance. They are asked to give a score of 1 to 10 points. For these five activities, they are also asked to score their satisfaction levels. In the same way, they give themselves points between 1 and 10 points (1: I am not satisfied at all, 10: I can be satisfied). Scores obtained from individuals about both performance and satisfaction levels are collected separately and divided by the number of activities. Average scores related to performance and satisfaction are determined.

CONTACTS AND LOCATIONS:
Overall Officials: FERRUH TAŞPINAR, Prof. Dr., Principal Investigator — Izmir Democracy University
Locations (1):
- Betül TAŞPINAR, Konak, İ̇zmi̇r, Turkey (Türkiye)